CLINICAL TRIAL: NCT06932393
Title: A Randomized, Double-blind, Single-center, Self-controlled Exploratory Clinical Study of Exosomes for Hairloss Treatment
Brief Title: Exosomes for Hairloss Treatment
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Guangzhou Bio-gene Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BG-CT-24-007
Record Dates: First submitted 2025-04-09; First posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Hair Loss
Keywords: Hair Loss; Exosomes
MeSH Terms: conditions — Alopecia | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- exosomes (Experimental): Subjects will receive 5E8 ~5E9 particles/cm² of exosome therapy in the study area during the dose escalation phase.
  Interventions: Biological: exosomes
- saline (Placebo Comparator): The control site will receive the same volume of saline as the exosomes administered in the study site.
  Interventions: Other: saline

INTERVENTIONS:
Biological: exosomes — Each subject will receive 3 injections with an interval of one month.
  Other Names: EVs
  Arms: exosomes
Other: saline — Each subject will receive 3 injections with an interval of one month.
  Arms: saline

SUMMARY:
Many people suffer from alopecia, which is caused by hereditary factors, emotional stress, and psychiatric disorders. There are devastating physical and psychological consequences as a result. Exosomes are isolated from donated human mesenchymal stem cells and purified using specific processing. This study is a randomized, double-blind, dose-escalation clinical trial designed to evaluate the efficacy and safety of exosomes therapy for alopecia.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects are able to read documents and can sign informed consent.
2. 18~75 years old (including the threshold), gender is not limited.
3. The subject's "hair loss grade" meets the following criteria:

1) BASP grade: Basic type (M2 to M3, or C2 to C3, or U1 to U3) or special type (V1 to V3, or F1 to F3); 2) For female: Ludwig Grade I to II. Or for male: Hamilton-Norwood Grade III to IV; 3) Hair density by phototrichogram: ≤ 190 hair/cm² ; 4. Hair dryness ≥ 5%; 5. Until withdrawal/completion of the study, subjects agree not to undergo any topical treatment for hair loss and agree to use a neutral shampoo.

Exclusion Criteria:

1. People with patchy or diffuse baldness, syphilitic alopecia, scarring alopecia, malnutrition, chemotherapy/radiotherapy-induced hair loss.
2. Those with a combination of diseases that have an impact on hair growth.
3. Use of medications, medicated shampoos, or hair care products that may interfere with efficacy evaluation within 3 months prior to screening (oral administration of therapeutic agents for androgenetic alopecia must be discontinued for at least 6 months).
4. Have received scalp radiation and/or laser or surgical therapy within 3 months prior to screening.
5. Participated or are participating in a interventional clinical trial within 3 months.
6. Persons with a history of hereditary alopecia areata.
7. Women who are pregnant or breastfeeding, or male/female subjects whose own/partner's pregnancy is planned within 6 months.
8. Have undergone hair transplantation in the previous 24 months.
9. Individuals testing positive for active infectious diseases or carriers of communicable pathogens.
10. Those with keloid, keloid-prone or hyperplastic scarring.
11. Those who, in the opinion of the investigator, are otherwise unfit to participate in this clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-04-30 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Comparison of localized hair density | 3rd month after 3 treatments
  Quantify hair counts within designated 1.5 cm × 1.5 cm fixed areas in both the study area and control area, and compare the localized hair density (hair/cm²) between the two areas.
Safety Assessment | From the initial treatment administration to the subject withdrawal from the study.
  Incidence of treatment emergent adverse events (TEAEs)
Comparison of overall hair density | 3rd month after 3 treatments
  Evaluate and score overall hair density in both the study area and control area using an 8-level assessment scale, followed by a comparative analysis of the two areas.

SECONDARY OUTCOMES:
Change of hair density | 3rd and 6st month after 3 treatments
  Change in hair density of study area with the baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen Qianhai Shekou Free Trade Zone Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided